CLINICAL TRIAL: NCT03507127
Title: Targeted Pharmacological and Behavioral Treatments for Smoking in Schizophrenia Study 1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low rate of enrollment
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Jennifer Tidey, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R21DA041114 (NIH)
Record Dates: First submitted 2018-04-05; First posted 2018-04-24 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Varenicline (Active Comparator)
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Standard dosing: 0.5 mg/day on days 1-3, 0.5 mg twice daily (morning, evening) on days 4-7, then 1 mg twice daily to the end of the medication period.
  Arms: Varenicline
Drug: Placebo — Dosing schedule matched to active comparator: on tablet on days 1-3, one tablet twice daily (morning, evening) on days 4-7, then one tablet twice daily to the end of the medication period.
  Arms: Placebo

SUMMARY:
Schizophrenia is associated with high rates of cigarette smoking and associated morbidity and mortality. In this study, smokers with schizophrenia will complete a baseline session and then randomized to varenicline (VAR) or placebo (PLA). After 1 week on medication, participants will complete a cigarette rating task session. Participants will then undergo a 72-hr abstinence period in which they will come to the laboratory twice per day and receive high-value cash reinforcement contingent upon meeting a strict breath CO abstinence criterion. At each visit, they will rate withdrawal symptoms, mood and craving. At the end of the abstinence period, they will repeat the cigarette rating task. Participants will return to the lab to provide a CO sample 24 hours later, and will text the lab with videos of their CO samples for one week. Date and time of smoking relapse will be measured from these samples.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women
2. Ages 18-65
3. Have schizophrenia or schizoaffective disorder
4. Would like to quit smoking within the next 6 months
5. Have smoked at least 10 cigarettes per day in the past year
6. Have breath CO level > 10 ppm
7. Able to speak, read and comprehend English well enough to complete study procedures

Exclusion Criteria:

1. Pregnant, breast-feeding, or unwilling to use medically-approved contraception
2. Currently using varenicline, bupropion or nicotine replacement therapy for smoking cessation
3. Medical disease that would preclude participation
4. Unstable psychiatric conditions
5. Body mass index (BMI) < 15 or > 38 kg/m2
6. Past-month suicidal intention, with or without a specific plan
7. Positive urine drug screen or breath alcohol level > 0.01% at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gender is based on self-report
Enrollment: 5 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tidey, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, 121 South Main Street, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 3 | 2
Completed | 1 | 1
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Unable to meet smoking abstinence criterion | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (8.5) | 46 (7.1) | 50 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Fagerstrom Test of Nicotine Dependence score [Mean (Standard Deviation); unit: units on a scale] — This scale measures nicotine dependence severity. Total score is reported, and scores can range from 0-10, with higher scores indicating more severe dependence.
  units on a scale | 8.3 (2.1) | 6.5 (0.7) | 7.6 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Questionnaire on Smoking Urges - Brief Form
Description: Average of all items, rated from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate higher levels of smoking urge or craving.
Time Frame: 72 hrs abstinence
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 3 | 2
score on a scale | 3.12 (2.11) | 4.41 (2.72)

2. Primary Outcome: Minnesota Nicotine Withdrawal Scale - Negative Affect Scale
Description: Average of responses to the anger, depression, anxiety and difficulty concentrating items, which are rated from 0 (not present) to 4 (severe).
Time Frame: 72 hrs abstinence
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 3 | 2
score on a scale | 1.45 (0.57) | 0.85 (0.92)

3. Secondary Outcome: Modified Cigarette Evaluation Questionnaire - Satisfaction Scale
Description: Average of the satisfaction, taste and enjoyment items, which are rated from 1 (not at all) to 7 (extremely)
Time Frame: 72 hrs abstinence
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 3 | 2
score on a scale | 5.33 (1.15) | 3.43 (1.20)

4. Secondary Outcome: Modified Cigarette Evaluation Questionnaire - Reward Scale
Description: Average of the calm, feel more awake, less irritable, help to concentrate and reduce hunger items, which are rated from 1 (not at all) to 7 (extremely)
Time Frame: 72 hrs abstinence
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 3 | 2
score on a scale | 4.00 (0.35) | 4.30 (0.0)

5. Secondary Outcome: Latency to Smoking Relapse
Description: hours until relapse during a smoking abstinence period, verified with breath carbon monoxide (CO) levels
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 1 | 1
hours | 8 (0) | 24 (0)

6. Other Pre Specified Outcome: Brief Psychiatric Rating Scale
Description: Sum of all items rated from 1 (not present) to 7 (extremely severe)
Time Frame: 72 hrs abstinence
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 3 | 2
score on a scale | 1.33 (0.11) | 1.37 (0.06)

ADVERSE EVENTS:
Time Frame: 19 days
Arm/Group | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/2
Other Adverse Events (participants affected / at risk) | 1/3 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=3) | Placebo (N=2)
voluntary psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — Participant used alcohol and drugs leading to auditory hallucinations and voluntary psychiatric hospitalization. Determined to be unrelated to study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=3) | Placebo (N=2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — One participant experienced mild nausea and one instance of vomiting while in the study. The study physician reviewed these events and determined that they were expected, possibly related, and did not involve risk.

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT03507127/Prot_SAP_000.pdf